CLINICAL TRIAL: NCT00891644
Title: HIV-Related Care Engagement: Linkage to Care and Care-Seeking for HIV-Infected Adolescents, Phase II
Brief Title: Linkage to Care - Part II
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: ATN 066b
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-02

CONDITIONS: HIV; Care-seeking; HIV Infections
Keywords: HIV; Care-seeking
MeSH Terms: conditions — HIV Infections | interventions — Case Management

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: HIV positive adolescents who never initiated care within 6 months of receipt of HIV positive results.
  Interventions: Other: Case Management; Other: Snowball sampling
- 2: HIV positive adolescents who initiated care, but did not follow up with care within 12 months of the initial care visit. Also included in this group are those who initiated and followed-up with care, but have dropped out of care for 12 or more months.
  Interventions: Other: Referral Lists
- 3: HIV positive adolescents who initiated care and maintained care. These youth are currently in care.

INTERVENTIONS:
Other: Case Management — Clinical personnel at each AMTU site may work with other personnel from organizations authorized to have access to personal health information to identify clients identified as HIV positive within the past 6 - 18 months.
  Initial contact will be made by persons at source organizations who are authorized to have access to personal health information. Persons so authorized will explain the nature of the research study and request permission from the client for subsequent contact by research personnel from the AMTU site. If permission for contact is received, research personnel at each site will attempt calls as specified by the potential participant or at random times (before 12:00 pm; between 12:00 - 4:00 pm; and between 4:00 - 10:00 pm) for no more than 10 attempts.
  Groups: 1
Other: Snowball sampling — Snowball sampling assumes that social networks of HIV sero-positive persons in treatment may overlap with those of HIV sero-positive persons not in treatment.
  When a site is assigned to identify HIV positive adolescents not in care by snowball sampling, all HIV positive persons in care at the site will be invited to refer other adolescents known to them as HIV positive, but not in care, for possible participation in the study.
  Printed information containing a brief description of the research in English and in Spanish and contact information of site study personnel will be provided to in-care adolescents at the site for distribution to those known HIV positive adolescents who are not in care.
  Groups: 1
Other: Referral Lists — AMTU staff will develop lists of potential participants at their sites who have had an initial HIV-related health care visit but not received additional visits within the 12 mos prior the list (or before protocol screening) or have completed initial and follow up visits but dropped out of care for 12 or more mos. Back-up lists will be made of potential participants who have gone 9-12 mos and 6-9 mos without a visit. Clinical staff at each AMTU may work with staff from other organizations authorized to access personal health information to find potential participants. 1st contact will be made by persons at source organizations who are authorized to access personal health information. Authorized staff will explain the study and ask permission for contact by research staff at the AMTU site. If so, research staff will attempt calls as specified by the potential participant or at random (before 12 pm; between 12-4 pm; and between 4-10 pm) for no more than 10 attempts.
  Groups: 2

SUMMARY:
This is the second phase of a two-phase, cross-sectional study of linkage to medical care of HIV positive youth. Social, psychological and behavioral factors associated with receipt of care will be evaluated. This study will also compare three methods for recruitment of out-of-care youth using a randomized permuted block list of possible sequences.

DETAILED DESCRIPTION:
ATN 066b consists of a cross-sectional evaluation of three groups of recently diagnosed HIV-infected adolescents including: (1) care non-initiation; (2) care initiation, no maintenance; and (3) care initiation with maintenance. Social, psychological and behavioral factors associated with HIV-related care-seeking will be assessed using an ACASI. Three recruitment strategies using a randomized permuted block list of possible sequences for HIV-infected youth not in care will be also compared.

The ACASI instrument will be adapted from previously used instruments intended to retrospectively reconstruct the care-seeking process and to assess quality of life, concerns and expectations for care, satisfaction with care, and social-problem solving.

Ideally, the ACASI will be administered during a single session and may take up to 90 minutes to complete. Participants who are unable to complete the ACASI in one session will be allowed up to 7 days after initiation to complete it. Completion of all study data collection, including accrual period, is expected to take approximately 12 months. Outcome measures will be classified as (1) care non-initiation; (2) care initiation, no maintenance; or (3) care initiation and maintenance.

The assessment of recruitment strategies most effective for not in care youth will include: use of usual case-management approaches; snowball sampling and venue-based advertisement.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection behaviorally-acquired at age 10 years or older, by the site staff's best determination;
* HIV-1 infection documented by a positive result on any of the following licensed tests at any time: any HIV-1 antibody test confirmed by Western blot, HIV-1 culture, HIV-1 DNA PCR, or plasma HIV-1 RNA PCR > 1,000 copies/ml; NOTE: Anonymous HIV-1 antibody test results, with confirmation by Western blot, will be considered an acceptable form of documentation for those individuals who do not wish to have their name linked to their HIV diagnosis. The original slip containing the result will need to be presented. If individuals request that their test results remain anonymous, AMTUs are encouraged to retest using an anonymous method.
* Documented or self-reported receipt of HIV positive diagnosis between 6 -18 months, inclusive, prior to the protocol screening date; NOTE: The protocol team will monitor enrollment during the first 3 months of study implementation and may expand this window to 24 months, if necessary.
* Ages 14 - 24 years, inclusive at the time of protocol screening;
* Ability to understand and willingness to provide written informed consent/assent in English or Spanish;
* Group 1: Never initiated HIV-related medical care and 6 or more months have elapsed since receipt of an HIV diagnosis. This cohort is not currently considered in care;
* Group 2: Initiated HIV-related medical care, but 12 or more months have elapsed since care was initiated, and has not had additional HIV-related medical care since the initial visit; or
* Group 2: Initiated and had follow up HIV-related medical care, but is no longer in care for 12 or more months since the last visit. This cohort is not currently considered in care; and
* Group 3: Initiated and maintained HIV-related medical care with at least one maintenance visit within the 12 months prior to the protocol screening date. This cohort is currently considered in care.

Exclusion Criteria:

* Psychiatric disorder (untreated) associated with thought disorder, hallucinations, acute substance use withdrawal. Stabilized patients receiving appropriate psychiatric care will not be excluded if informed consent can be reasonably assumed;
* Visibly distraught and/or visibly emotionally unstable (e.g., depressive mood; exhibiting manic, suicidal, or violent behavior);
* Active drug or alcohol use or dependence that, in the opinion of the site personnel, would interfere with ability to give true informed consent and to adhere to the study requirements;
* Known pregnancy;
* Acute illness that, in the opinion of the treating clinician, would endanger the well-being of the individual if treatment was delayed due to study participation;
* HIV positive adolescents infected through either perinatal transmission or blood products, including those who became aware of their HIV diagnosis within the prior 6 -18 months; and
* Explicit prior refusal of permission by the adolescent for any subsequent contact by site personnel. (Adolescents who wish to participate and provide signed informed consent, but who cannot or will not provide contact information, do not meet this exclusion criterion.)

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 1. Behaviorally-infected, HIV positive adolescents, informed of their HIV diagnosis within 6-18 months of the protocol screening date, who provide consent for study participation;
  2. Ages 14-24 years, inclusive at the time of protocol screening;
  3. Males and females; and
  4. English- or Spanish-speaking
  Group 1 - HIV positive adolescents who never initiated care within 6 months of receipt of HIV positive results; Group 2 - HIV positive adolescents who initiated care, but did not follow up with care within 12 months of the initial care visit. Also included in this group are those who initiated and followed-up with care, but have dropped out of care for 12 or more months; and Group 3 - HIV positive adolescents who initiated care and maintained care. These youth are currently in care.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2009-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Retrospectively recreate the process and timeline of care-seeking among screened HIV positive adolescents. | 1 year

SECONDARY OUTCOMES:
Evaluate technical aspects of identification and recruitment of HIV positive adolescents who have not engaged in care or who have not maintained care. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Fortenberry, MD, Study Chair — Adolescent Trials Network
Locations (5):
- United States (5):
  - Children's Hopsital of Los Angeles, Los Angeles, California
  - Children's Diagnostic and Treatment Center, Fort Lauderdale, Florida
  - Childrens Memorial Hospital, Chicago, Illinois
  - Children's Hospital at Montefiore Medical Center, The Bronx, New York
  - Children's Hopsital of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- See also: ATN Website — https://www.atnonline.org